CLINICAL TRIAL: NCT07232693
Title: The Impact of Home-Based Telerehabilitation Versus Center-Based Cardiac Rehabilitation on Anxiety, Depression, and Quality of Life After Coronary Artery Bypass Grafting: A Randomized Controlled Trial
Brief Title: Telerehabilitation vs. Center-Based Rehab for Psychological Well-being After CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yan Liu, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S00775-2
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Psychological Distress After Coronary Artery Bypass Grafting (CABG)
Keywords: Coronary Artery Bypass Grafting; Telerehabilitation; Anxiety; Depression; Quality of Life; Cardiac Rehabilitation
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home-Based Telerehabilitation (HBTCR) Group (Experimental): Participants received a personalized 12-week exercise program to perform at home. They were provided with a wearable heart rate monitor and a mobile application to log their activities. A dedicated cardiac rehabilitation nurse contacted each patient weekly via phone or video call to review progress, adjust the exercise plan, and provide structured psychosocial support and counseling.
  Interventions: Behavioral: Home-Based Telerehabilitation Cardiac Rehabilitation
- Center-Based Cardiac Rehabilitation (CBCR) Group (Active Comparator): Participants attended 36 supervised sessions at the hospital's cardiac rehabilitation center over 12 weeks (3 sessions/week). Each session included aerobic and resistance exercises. In addition, patients attended weekly group sessions for health education and psychosocial support, covering topics like stress management and coping strategies.
  Interventions: Behavioral: Home-Based Telerehabilitation Cardiac Rehabilitation
- Control Group (Sham Comparator): Participants received usual care, which included standard postoperative medical advice and health education pamphlets detailing general recommendations for diet, medication, and physical activity. They did not receive any structured exercise prescription or formal psychological support from the study team.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Home-Based Telerehabilitation Cardiac Rehabilitation — A 12-week structured and remotely monitored cardiac rehabilitation program including a personalized exercise prescription (aerobic and resistance training), remote monitoring with a wearable heart rate sensor and mobile app, and weekly one-on-one psychosocial support and counseling via phone or video call from a rehabilitation nurse.
  Arms: Home-Based Telerehabilitation (HBTCR) Group
Behavioral: Home-Based Telerehabilitation Cardiac Rehabilitation — A 12-week structured and remotely monitored cardiac rehabilitation program including a personalized exercise prescription (aerobic and resistance training), remote monitoring with a wearable heart rate sensor and mobile app, and weekly one-on-one psychosocial support and counseling via phone or video call from a rehabilitation nurse.
  Arms: Center-Based Cardiac Rehabilitation (CBCR) Group
Behavioral: Usual Care — Standard postoperative care including prescribed medications and routine follow-up, supplemented with health education pamphlets on lifestyle modification. No structured or supervised rehabilitation was provided.
  Arms: Control Group

SUMMARY:
This randomized controlled trial aims to determine if a 12-week home-based telerehabilitation (HBTCR) program is as effective as traditional center-based cardiac rehabilitation (CBCR) in improving psychological well-being (anxiety and depression) and quality of life in patients who have undergone coronary artery bypass grafting (CABG). A third group receiving usual care served as a control.

DETAILED DESCRIPTION:
Psychological distress, such as anxiety and depression, is common after coronary artery bypass grafting (CABG) and negatively affects recovery and quality of life. While center-based cardiac rehabilitation (CBCR) effectively addresses these issues, participation is often limited by barriers like travel, cost, and scheduling. Home-based telerehabilitation (HBTCR) offers a potential solution. This single-center, prospective, three-arm randomized controlled trial was designed to compare the effectiveness of HBTCR versus CBCR and usual care. A total of 110 clinically stable patients, 4-8 weeks post-CABG, were randomly assigned in a 1:1:1 ratio to an HBTCR group, a CBCR group, or a control group. The intervention period was 12 weeks. The study hypothesized that the HBTCR program, which includes a personalized exercise plan, remote monitoring via a wearable device and mobile app, and weekly psychosocial support from a nurse, would be as effective as the traditional supervised in-person CBCR program in reducing symptoms of anxiety and depression and improving health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-75 years.
* 4-8 weeks post-Coronary Artery Bypass Grafting (CABG).
* In clinically stable condition.
* Had access to a smartphone and were willing to use it for the program.
* Willing to participate in a 12-week rehabilitation program.
* Provided written informed consent.

Exclusion Criteria:

* Presence of severe and unstable comorbidities (e.g., uncontrolled heart failure, recent stroke).
* Severe orthopedic limitations that would prevent participation in exercise.
* Significant cognitive impairment or psychiatric disorders that would interfere with participation.
* Inability to provide informed consent.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety Symptoms | Baseline, 12 Weeks
  The change from baseline in the Hamilton Anxiety Scale (HAMA) score. The HAMA scale is a clinician-rated scale where higher scores indicate greater symptom severity.
Change in Depression Symptoms | Baseline, 12 Weeks
  The change from baseline in the 17-item Hamilton Depression Scale (HAMD) score. The HAMD is a clinician-rated scale where higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Change in Health-Related Quality of Life | Baseline, 12 Weeks
  The change from baseline in scores on the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36). The SF-36 assesses eight domains: Physical Functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role-Emotional (RE), and Mental Health (MH). Scores for each domain range from 0 to 100, with higher scores indicating better quality of life.

OTHER OUTCOMES:
Change in Peak Oxygen Consumption (VO₂ peak) | Baseline, 12 Weeks
  The change from baseline in VO₂ peak, a measure of cardiopulmonary fitness, assessed via an exercise test. Unit: mL/kg/min.
Change in 6-Minute Walk Distance (6MWD) | Baseline, 12 Weeks
  The change from baseline in the distance a patient can walk in six minutes, measuring functional exercise capacity. Unit: Meters.
Change in Left Ventricular Ejection Fraction (LVEF) | Baseline, 12 Weeks
  The change from baseline in LVEF, assessed by echocardiography. Unit: Percentage (%).
Adherence Rate | Through study completion, 12 weeks
  The percentage of completed cardiac rehabilitation sessions out of the total prescribed sessions for the HBTCR and CBCR groups.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China